CLINICAL TRIAL: NCT01205048
Title: A Pivotal USA Randomized, Evaluator-blinded, Active-controlled, Multi-center, Split-face Comparison Study of Emervel Classic Lidocaine Versus Juvederm® Ultra in the Treatment of Moderate to Severe Facial Wrinkle Folds
Brief Title: Emervel Classic Lidocaine Versus Juvederm® Ultra in Treatment of Moderate to Severe Facial Wrinkles and Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.06.CIP.18156
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Skin Wrinkling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emervel Classic Lidocaine (Experimental): NLFs (Nasolabial Folds) were injected with Emervel Classic Lidocaine (20 mg/mL with 0.3% lidocaine).
  Interventions: Device: Emervel Classic Lidocaine
- Juvederm® Ultra (Active Comparator): NLFs were injected with Juvéderm Ultra (24 mg/mL).
  Interventions: Device: Juvederm® Ultra

INTERVENTIONS:
Device: Emervel Classic Lidocaine — 20 mg/mL + 0.3% lidocaine
  Arms: Emervel Classic Lidocaine
Device: Juvederm® Ultra — 24mg/mL
  Arms: Juvederm® Ultra

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of Emervel Classic Lidocaine versus Juvederm® Ultra in the treatment of moderate to severe facial wrinkles and folds.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female 18 years of age or older
* The subject has bilateral nasolabial folds that, in the opinion of both the Blinded Evaluating Investigator and the Unblinded Injecting Investigator, can be corrected with an injectable dermal implant
* The subject has the same Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 (moderate or severe) for each nasolabial fold

Exclusion Criteria:

* The subject has active skin disease or inflammation on or near a nasolabial fold that, in the Principal Investigator's opinion, would interfere with the study device injections and/or study assessments.
* The subject has a history of sensitivity to hyaluronic acid
* The subject has a history of sensitivity to lidocaine or other amide type anesthetics
* The subject is, in the Principal Investigator's opinion, at undue risk based on the precautions, warnings and contraindications for local lidocaine anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2011-06-27 (Actual); Study Completion 2012-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Chair — Galderma R&D
Locations (12):
- United States (12):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Skin Care & Laser Physicians of Beverly Hills, Los Angeles, California
  - FacesPlus Aesthetic Facility, San Diego, California
  - Therapeutics Research, San Diego, California
  - Steven Fagien, Boca Raton, Florida
  - Dermatology Research Institute, Coral Gables, Florida
  - Laser & Skin Surgery Center in Indiana, Carmel, Indiana
  - Callender Center for Clinical Research, Glendale, Maryland
  - The Center for Dermatology, Cosmetic & Laser Surgery, Mount Kisco, New York
  - Sadick Research Group, New York, New York
  - Oregon Medical Research PC, Portland, Oregon
  - DermResearch, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 centers in the United States from September 2010 to January 2012.
Pre-assignment Details: A total of 171 participants were enrolled, of which 170 participants received treatment in this study.
Groups:
- All Participants: Participants were randomized to receive either Emervel Classic Lidocaine (20 milligram per milliliter [mg/mL] with 0.3% lidocaine) injection in the left nasolabial fold (NLF) and Juvederm Ultra (24 mg/mL) injection in to the right NLF or Juvederm Ultra (24 mg/mL) injection in the left NLF and Emervel Classic Lidocaine (20 mg/mL with 0.3% lidocaine) injection in the right NLF.
Period: Overall Study
Arm/Group | All Participants
Started | 170
Emervel Classic Lidocaine in Left NLF Followed by Juvederm Ultra in Right NLF | 84
Juvederm Ultra in Left NLF Followed by Emervel Classic Lidocaine in Right NLF | 86
Completed | 149
Not Completed | 21
Not completed — Withdrawal by Subject | 14
Not completed — Clinical Investigation Plan Violation | 1
Not completed — Lost to Follow-up | 4
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: The Intent to treat (ITT) population was defined as all participants who were randomized and received an injection on both treatment sides.
Groups:
- Emervel Classic Lidocaine in Left NLF Followed by Juvederm Ultra in Right NLF: Participants received Emervel Classic Lidocaine (20 mg/mL with 0.3% lidocaine) injection into the left NLF and Juvéderm Ultra (24 mg/mL) in the right NLF.
- Juvederm Ultra in Left NLF Followed by Emervel Classic Lidocaine in Right NLF: Participants received Juvéderm Ultra (24 mg/mL) injection into the left NLF and Emervel Classic Lidocaine (20 mg/mL with 0.3% lidocaine) injection in the right NLF.
- Total: Total of all reporting groups
Arm/Group | Emervel Classic Lidocaine in Left NLF Followed by Juvederm Ultra in Right NLF | Juvederm Ultra in Left NLF Followed by Emervel Classic Lidocaine in Right NLF | Total
Number analyzed (Participants) | 84 | 86 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.82) | 53.6 (7.64) | 53.9 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 81 | 160
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 58 | 58 | 116
  Black | 5 | 10 | 15
  Hispanic | 20 | 18 | 38
  Other | 1 | 0 | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  Participants
    Skin Type I | 3 | 3 | 6
    Skin Type II | 19 | 20 | 39
    Skin Type III | 29 | 23 | 52
    Skin Type IV | 27 | 28 | 55
    Skin Type V | 4 | 5 | 9
    Skin Type VI | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Scale (WSRS) at Week 24 After Final Initial Injection
Description: WSRS is a validated 5-point reference scale with photographs that classifies facial wrinkles (nasolabial folds). WSRS represents clinically meaningful change in NLF severity from the adjacent grades where 1= absent (no visible fold; continuous skin line), 2 = mild (shallow but visible fold with a slight indentation; minor facial feature; implant expected to produce a slight improvement in appearance), 3 = excellent (correction is expected from injectable implant), 4 = severe (very long and deep folds; prominent facial feature; less than 2 mm visible fold when stretched; significant improvement expected from injectable implant), 5 = extreme (extremely deep and long folds, detrimental to facial appearance; 2 to 4 millimeter (mm) visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 24 after final initial injection
Population: Intent to Treat (ITT) population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Emervel Classic Lidocaine: NLFs were injected with Emervel Classic Lidocaine (20 mg/mL with 0.3% lidocaine).
- Juvederm Ultra: NLFs were injected with Juvéderm Ultra (24 mg/mL).
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Score on a scale | -1.1 (0.75) | -1.2 (0.76)

2. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Scale (WSRS) at Week 3 After the Final Initial Injection
Description: WSRS is a validated 5-point reference scale with photographs that classifies facial wrinkles (nasolabial folds). WSRS represents a clinically meaningful change in NLF severity from the adjacent grades where 1 = absent (no visible fold; continuous skin line), 2 = mild (shallow but visible fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance), 3 = excellent (correction is expected from injectable implant), 4 = severe (very long and deep folds; prominent facial feature; less than 2 mm visible fold when stretched; significant improvement is expected from injectable implant), 5 = extreme (extremely deep and long folds, detrimental to facial appearance; 2 to 4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 3 after final initial injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Score on a scale | -1.7 (0.72) | -1.8 (0.70)

3. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Scale (WSRS) at Week 12 After Final Initial Injection
Description: WSRS is a validated 5-point reference scale with photographs that classifies facial wrinkles (nasolabial folds). WSRS represents a clinically meaningful change in nasolabial fold severity from the adjacent grades where 1 = absent (no visible fold; continuous skin line), 2 = mild (shallow but visible fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance), 3 = excellent (correction is expected from injectable implant), 4 = severe (very long and deep folds; prominent facial feature; less than 2 mm visible fold when stretched; significant improvement is expected from injectable implant), 5 = extreme (extremely deep and long folds, detrimental to facial appearance; 2 to 4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12 after final initial injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
score on a scale | -1.5 (0.75) | -1.5 (0.78)

4. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Scale (WSRS) at Week 36 After Final Initial Injection
Description: as for outcome 2
Time Frame: Baseline, Week 36 after final initial injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Score on a scale | -1.0 (0.75) | -1.1 (0.74)

5. Secondary Outcome: Mean Change From Baseline in Wrinkle Severity Rating Scale (WSRS) at Week 48 After Final Initial Injection
Description: as for outcome 2
Time Frame: Baseline, Week 48 after final initial injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Score on a scale | -0.7 (0.69) | -0.9 (0.76)

6. Secondary Outcome: Mean Change From Baseline in Participant Self-Assessment of Wrinkle Severity at Week 24 After Final Initial Injection
Description: Participants self-assessment was measured by using a wrinkle severity scale with 1 being absent and 5 being extreme. Each participant was to perform an assessment of the wrinkle severity based on self-assessment score: 1= Absent (No visible fold; continuous skin line), 2= Mild (Shallow but visible fold with a slight indentation), 3= Moderate (Moderately deep folds), 4= Severe (Very long and deep fold), 5= Extreme (Extremely deep and long folds). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 24 after final initial injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Score on a scale | -1.3 (1.04) | -1.4 (0.96)

7. Secondary Outcome: Participant Pain Assessment After the Initial Injection
Description: Participant pain severity for each NLF was assessed at time 0, 15, 30, 45, 60 minutes and 24 hours after the initial injection using an 11-point Numeric Pain Intensity Scale (NPIS).The NPIS was a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with 0 is no pain and 10 is the worst possible pain.
Time Frame: At 0 ,15, 30, 45, 60 minutes and 24 hours after the initial injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides. "Here, "number analyzed signifies who were evaluable at the given timepoints".
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Score on a scale
  At 0 Minutes | 2.9 [0 to 8] | 5.6 [0 to 10]
  At 15 Minutes | 0.5 [0 to 6] | 2.1 [0 to 8]
  At 30 Minutes | 0.2 [0 to 4] | 1.1 [0 to 8]
  At 45 Minutes | 0.2 [0 to 3] | 0.7 [0 to 7]
  At 60 Minutes | 0.1 [0 to 2] | 0.5 [0 to 5]
  At 24 Hours: number analyzed (Participants) | 168 | 168
  At 24 Hours | 0.4 [0 to 5] | 0.4 [0 to 4]

8. Secondary Outcome: Participant Pain Assessment After the Initial Touch-up Injection
Description: as for outcome 7
Time Frame: At 0, 15, 30, 45, 60 minutes and 24 hours after the Initial Touch-up Injection
Population: ITT population included participants who were randomized and received an injection on both treatment sides. "Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure and number analyzed signifies who were evaluable at the given timepoints.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 90 | 86
Score on a scale
  At 0 Minutes | 2.3 [0 to 8] | 4.4 [0 to 10]
  At 15 Minutes | 0.3 [0 to 4] | 1.4 [0 to 6]
  At 30 Minutes | 0.2 [0 to 3] | 0.6 [0 to 5]
  At 45 Minutes | 0.1 [0 to 2] | 0.3 [0 to 4]
  At 60 Minutes | 0.1 [0 to 2] | 0.2 [0 to 3]
  At 24 Hours: number analyzed (Participants) | 82 | 79
  At 24 Hours | 0.2 [0 to 2] | 0.3 [0 to 4]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the study drug. Number of participants with AEs were reported. Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Time Frame: From start of study drug administration up to 56 weeks
Population: The safety population included all participants who received at least one injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
Number analyzed (Participants) | 170 | 170
Participants | 66 | 64

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 56 weeks
Description: The safety population included all participants who received at least one injection.
Arm/Group | Emervel Classic Lidocaine | Juvederm Ultra
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/170
Serious Adverse Events (participants affected / at risk) | 2/170 | 2/170
Other Adverse Events (participants affected / at risk) | 10/170 | 11/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Emervel Classic Lidocaine (N=170) | Juvederm Ultra (N=170)
Cholecystitis (General disorders) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
Worsening right knee osteoarthritis (General disorders) | 1 | 1 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Emervel Classic Lidocaine (N=170) | Juvederm Ultra (N=170)
Headache (Nervous system disorders) | 10 | 11 — Event was unrelated to study product or injection procedure. If the treated side where an AE occurred was not applicable, this AE was summarized under each treatment group."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other